CLINICAL TRIAL: NCT02626611
Title: A Phase 2 Study Multi Oral Immunotherapy in Multi Food Allergic Patients to Test Tolerance M-TAX Study
Brief Title: Multi Immunotherapy to Test Tolerance and Xolair
Acronym: M-TAX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kari Christine Nadeau (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Children's Hospital of Philadelphia (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital Los Angeles (Other); University of Washington (Other)
Responsible Party: Sponsor-Investigator, Kari Christine Nadeau, Sponsor Investigator, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 28942
Record Dates: First submitted 2015-11-24; First posted 2015-12-10 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Food Allergy
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks. The oat placebo food, will be compared to high dose (2000 milligrams or low dose 300 milligrams food immunotherapy). At week 36 a food challenge will be performed to assess study endpoints.
  Interventions: Drug: Omalizumab; Drug: Food Flour Buildup
- Low Dose Food (Active Comparator): Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks. The oat placebo food, will be compared to high dose (2000 milligrams or low dose 300 milligrams food immunotherapy). At week 36 a food challenge will be performed to assess study endpoints.
  Interventions: Drug: Omalizumab; Drug: Food Flour Buildup
- High Dose Food (Active Comparator): Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks. The oat placebo food, will be compared to high dose (2000 milligrams or low dose 300 milligrams food immunotherapy). At week 36 a food challenge will be performed to assess study endpoints.
  Interventions: Drug: Omalizumab; Drug: Food Flour Buildup

INTERVENTIONS:
Drug: Omalizumab — Omalizumab is an anti-Immunoglobulin E antibody injection and will be administered per product insert from weeks 0 through 16 of the study.
  Other Names: Xolair
Drug: Food Flour Buildup — Food flours identified as allergic (based on food challenge), will be introduced at week 8. The food dose will be escalated every 2 weeks up to 2000 milligrams of each of the food flours. Subjects are required to reach 300 milligrams at week 16 to continue to week 30. Subjects must tolerate 2000 milligrams per food by week 28 in order to be randomized.

SUMMARY:
This is a phase 2 randomized, double-blind, placebo controlled study which will be conducted at multiple centers in the U.S. All subjects will receive oral immunotherapy for their specific food allergies (limited to 5 of those food allergens in Investigational New Drug (IND) 14831). All subjects will receive Omalizumab for 16 weeks. The subject's allergens will be introduced in a rush desensitization day at week 8. Subjects will return to clinic to escalate the dose of their allergens until 2,000mg protein of each allergen is reached Subjects will return to clinic for a DBPCFC to each allergen at week 30. If subjects are nonreactive to 2 or more allergens during their DBPCFC at week 30 they will be randomized to one of three double blinded arms: Arm A- continue with current dose (2000 mg each food allergen protein), Arm B-300 mg of each food allergen protein, Arm C-placebo (avoiding food allergen protein), their current dose. All subjects will return to clinic for a DBPCFC to each allergen at week 36. The final challenge of week 36 will be the final end of study visit.

Safety is a paramount concern in the study design and will be monitored carefully throughout the study. Study subjects and their parents/guardians will receive extensive education on food allergy reactions and medication use.

DETAILED DESCRIPTION:
The investigators will enroll multi food allergic subjects (4-55 years of age) with proven multi food allergies. The investigators anticipate enrolling 70 subjects with multi food allergies at more than one site. Subjects must have food specific Immunoglobulin E >4 kilo Units/Liter for each allergen or a skin test reactivity to each food allergen greater than or equal to 6mm wheal diameter. In addition, subjects must have a total Immunoglobulin E <2,000 kilo Units/Liter, a clinical reaction during a double blind placebo controlled food challenge (DBPCFC) with food protein/powder to establish sensitivity to given food protein/powder (pecan, milk, egg, peanut, almond, wheat, cashew, sesame seed, soy, walnut, hazelnut, shrimp, cod, salmon) and no clinical reaction during placebo (oat) as per Chemistry Manufacturing and Control section of Investigational New Drug.

Each subject is planned to be enrolled in the active phase of the study for 36 weeks.

Food protein and powder will be obtained and prepared as per Investigational New Drug 14831 and will be in compliance with all applicable regulations.

Omalizumab is approved by the European Medicines Agency (European FDA) for patients with severe asthma >6 years of age, and by the US FDA for patients >12 years of age. Omalizumab will be dosed according to Genentech Dosing Omalizumab will be provided by the site.

ELIGIBILITY:
Inclusion Criteria:

* Participant and/or parent guardian must be able to understand and provide informed consent and/or assent as applicable.
* Age 4 to 55 years with moderate to severe allergy to milk and/or egg and/or peanut and/or almond and/or wheat and/or cashew and/or sesame seed and/or soy and/or pecan and/or walnut and/or hazelnut
* Positive skin prick test result greater than or equal to 6 mm wheal diameter to each allergen OR
* ImmunoCAP Immunoglobulin E (IgE) level >4 kilo Unit/Liter for each allergen and
* A clinical reaction during a DBPCFC to small doses of food defined as < dose of 500 mg food protein
* No clinical reaction observed during the placebo (oat) challenge and
* If female, must have a negative urine pregnancy test on the same day (using a Clinical Laboratory Improvement Amendment (CLIA) approved urine test)
* If female, of child-bearing potential, must agree to be compliant with a medically-approved method of contraception (please see Pregnancy section under Patient Disposition in this protocol)
* Plan to remain in the study area of the research center during the trial
* Be trained on the proper use of the Epinephrine autoinjector
* Avoid open or blinded food challenges to other allergens outside this study

Exclusion Criteria:

* Inability or unwillingness of a participant/parent/guardian to give written informed consent or comply with study protocol
* History of cardiovascular disease
* History of other chronic disease (other than asthma, atopic dermatitis, or rhinitis) requiring therapy (e.g., heart disease, diabetes) that, in the opinion of the Principal Investigator, would represent a risk to the participant's health or safety in this study or the participant's ability to comply with the study protocol
* A total IgE at screening of >2,000 kU/L
* Previous adverse reaction to Xolair
* A history of severe anaphylaxis (defined as requiring intubation or admission to an ICU) to food allergens that will be used in this study
* Unstable angina, significant arrhythmia, uncontrolled hypertension, current smokers, chronic sinusitis, or other chronic or immunological diseases that, in the judgment of the investigator, might interfere with the evaluation or administration of the test drug or pose additional risk to the participant.
* Current use of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or betablockers (oral or topical)
* Routine use of medication that could induce adverse gastrointestinal reactions during the study
* Refusing to sign the Epinephrine autoinjector Training Form
* Pregnant or breast feeding women
* A history of oat allergy (since oat is the placebo agent in the DBPCFC), or an objective reaction to the screening DBPCFC to oat
* Unwilling to avoid all food allergen-containing items except those given as part of the Oral Immunotherapy as well as any other food allergens you are allergic to that are not included in the 10 foods listed in the study
* Concurrent/prior use of immunomodulatory therapy (within 1 month) ie, omalizumab, nontraditional forms of allergen immunotherapy (e.g., oral or sublingual)
* Severe asthma (2007 National Heart Lung and Blood Institute (NHLBI) Criteria Steps 5 or 6) at time of enrollment
* Mild or moderate asthma (2007 NHLBI Criteria Steps 1-4) at time of enrollment with any of the following criteria met:
* Forced Expiratory Volume at one second (FEV1) < 80% of predicted, or FEV1/Forced Vital Capacity (FVC) < 75%, with or without controller medications (only for age 6 or greater and able to do spirometry) or
* Inhaled Corticosteroid (ICS) dosing of > 220 mcg daily fluticasone (or equivalent inhaled corticosteroids based on NHLBI dosing chart) or
* 1 hospitalization in the past year for asthma or ER visit for asthma within the past six months
* Use of steroid medications (Intravenous (IV), Intramuscular (IM) or oral) in the following manners
* history of daily oral steroid dosing for >1 month during the past year or
* steroid burst course ( 5 or more days) of 1 mg/kg prednisone) course in the past 3 months or
* >2 steroid burst courses in the past year
* Use of complementary and alternative medicine (CAM) treatment modalities (e.g., herbal remedies) for atopic and/or non-atopic disease within 90 days preceding rush desensitization at week 8or at any time .
* Inability to discontinue antihistamines for the initial day of escalation, skin testing or Oral Food Challenges (OFCs)
* Use of investigational drugs within 24 weeks of participation
* Past or current medical problems or findings from physical assessment or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeau C Nadeau, MD PhD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Sean N. Parker Center for Allergy Research at Stanford University, Mountain View, California
  - Lurie Children's Hospital, Northwestern University, Chicago, Illinois
  - Mt. Sinai, Icahn School of Medicine, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Northwest Asthma & Allergy Center, Seattle, Washington

REFERENCES:
- [Derived] Andorf S, Purington N, Kumar D, Long A, O'Laughlin KL, Sicherer S, Sampson H, Cianferoni A, Whitehorn TB, Petroni D, Makhija M, Robison RG, Lierl M, Logsdon S, Desai M, Galli SJ, Rael E, Assa'ad A, Chinthrajah S, Pongracic J, Spergel JM, Tam J, Tilles S, Wang J, Nadeau K. A Phase 2 Randomized Controlled Multisite Study Using Omalizumab-facilitated Rapid Desensitization to Test Continued vs Discontinued Dosing in Multifood Allergic Individuals. EClinicalMedicine. 2019 Jan 21;7:27-38. doi: 10.1016/j.eclinm.2018.12.006. eCollection 2019 Jan. PMID 31193674

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants received Xolair but only those not withdrawn progressed to the Active Study Phase of allergen exposure.
Groups:
- Placebo; Low Dose Food: Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks. The oat placebo food, will be compared to high dose (2000 milligrams or low dose 300 milligrams food immunotherapy). At week 36 a food challenge will be performed to assess study endpoints.
  Omalizumab: Omalizumab is administered per product insert from weeks 0 -16 of the study.
  Food Flour Buildup: Food flours identified as allergic (based on food challenge), will be introduced at week 8. The food dose will be escalated every 2 weeks up to 2000 milligrams of each of the food flours. Subjects are required to reach 300 milligrams at week 16 to continue to week 30. Subjects must tolerate 2000 milligrams per food by week 28 in order to be randomized.
- High Dose Food: Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks. The oat placebo food, will be compared to high dose (2000 milligrams or low dose 300 milligrams food immunotherapy). At week 36 a food challenge will be performed to assess study endpoints.
  Omalizumab: Omalizumab is administered per product insert from weeks 0 - 16 of the study.
  Food Flour Buildup: Food flours identified as allergic (based on food challenge), will be introduced at week 8. The food dose will be escalated every 2 weeks up to 2000 milligrams of each of the food flours. Subjects are required to reach 300 milligrams at week 16 to continue to week 30. Subjects must tolerate 2000 milligrams per food by week 28 in order to be randomized.
Period: Overall Study
Arm/Group | Placebo | Low Dose Food | High Dose Food
Started | 20 | 21 | 19
Completed | 16 | 20 | 16
Not Completed | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Active phase (allergen exposure) participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Food | High Dose Food | Total
Number analyzed (Participants) | 20 | 21 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (4.9) | 8.1 (5.9) | 8.9 (3.2) | 9.3 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 3 | 23
  Male | 10 | 11 | 16 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 2 | 5
  White | 9 | 10 | 11 | 30
  More than one race | 2 | 3 | 1 | 6
  Unknown or Not Reported | 6 | 3 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 19 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Able to Tolerate an Oral Food Challenge to 2,000 mg at Least of 2 Allergens at Week 36 (i.e. the End of the Randomized Withdrawal/Tolerance Phase), Will be Reported.
Description: Number of FA participants who pass a DBPCFC to 2,000 mg each of 2 allergens (i.e. no reaction of grade 1 or more according to Bock's criteria) at week 36, will be reported.
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose Food | High Dose Food
Number analyzed (Participants) | 20 | 21 | 19
Participants | 11 | 17 | 17

2. Secondary Outcome: The Number of Participants Able to Tolerate an Oral Dose of 4,000mg Each of 2 Allergens Separately at Week 36, Will be Reported.
Description: Number of FA participants who pass a DBPCFC to (4,000 mg each of 2 allergens at week 36) (i.e. no reaction of grade 1 or more according to Bock's criteria) .
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Placebo; Low Dose Food; High Dose Food: Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food. At week 30, the cohort will be randomized into 3 groups (placebo, low dose food, and high dose food). Participants will continue on this dose for 6 weeks.
  Omalizumab: Omalizumab is an anti-Immunoglobulin E antibody injection and will be administered per product insert from weeks 0 through 16 of the study.
  Food Flour Buildup: Food flours identified as allergic (based on food challenge), will be introduced at week 8. The food dose will be escalated every 2 weeks up to 2000 milligrams of each of the food flours. Subjects are required to reach 300 milligrams at week 16 to continue to week 30. Subjects must tolerate 2000 m
Arm/Group | Placebo | Low Dose Food | High Dose Food
Number analyzed (Participants) | 20 | 21 | 19
Participants | 11 | 17 | 17

3. Secondary Outcome: The Number of Participants Able to Tolerate an Oral Dose of 2,000mg Each of 3 Allergens (When Applicable) Separately at Week 36, Will be Reported.
Description: Number of FA participants who pass a DBPCFC to 2,000 mg each of 3 allergens (when applicable) (i.e. no reaction of grade 1 or more according to Bock's criteria) at week 36, will be reported.
Time Frame: 36 weeks
Population: Number of participants analyzed reflects only those participants with 3 or more food allergies.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo; Low Dose Food; High Dose Food: Xolair will be administered in week 0 through 16 of the study. Starting at week 8, food doses will be serially increased, per protocol, to up to 2000 milligrams per food.
Arm/Group | Placebo | Low Dose Food | High Dose Food
Number analyzed (Participants) | 16 | 12 | 14
Participants | 8 | 12 | 13

4. Secondary Outcome: The Number of Participants Able to Tolerate an Oral Dose of 2,000mg Each of 4 Allergens (When Applicable) Separately at Week 36, Will be Reported.
Description: Number of FA participants who pass a DBPCFC to 2,000 mg each of 4 allergens (when applicable) (i.e. no reaction of grade 1 or more according to Bock's criteria) at week 36, will be reported.
Time Frame: 36 weeks
Population: Number of participants analyzed reflects only those participants with 4 or more food allergies
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose Food | High Dose Food
Number analyzed (Participants) | 9 | 10 | 8
Participants | 3 | 8 | 7

5. Secondary Outcome: The Number of Participants Able to Tolerate an Oral Dose of 2,000mg Each of 5 Allergens (When Applicable) Separately at Week 36, Will be Reported.
Description: Number of FA participants who pass a DBPCFC to 2,000 mg each of 5 allergens (when applicable) (i.e. no reaction of grade 1 or more according to Bock's criteria) at week 36, will be reported.
Time Frame: 36 weeks
Population: Number of participants analyzed reflects only those participants with 5 or more food allergies
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Low Dose Food | High Dose Food
Number analyzed (Participants) | 3 | 6 | 5
Participants | 0 | 5 | 5

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- All Participants Prior to Active Phase: Only Xolair administered before active phase began.
Arm/Group | All Participants Prior to Active Phase | Placebo | Low Dose Food | High Dose Food
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/20 | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/20 | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/70 | 0/20 | 0/21 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants Prior to Active Phase (N=70) | Placebo (N=20) | Low Dose Food (N=21) | High Dose Food (N=19)
abdominal pain (Gastrointestinal disorders) | 1 | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No